CLINICAL TRIAL: NCT05884203
Title: Improving Prosthetic Provision in Rural Communities: Limb Scanning With Caregiver Assistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F4276-R; I01RX004276 (NIH); 1676634 (Other: gov.irbnet.org)
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lower Extremity Amputation
Keywords: lower limb amputation; transtibial amputation; below knee amputation; prosthetic socket; prosthesis

STUDY DESIGN:
Intervention Model Description: The shape of the participants' residual limb will be captured with both study helper assistance and digital methods, and also by a prosthetist using traditional methods. However, only one study socket, randomly assigned, will be manufactured and used for outcomes testing.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants: Subjects will be blinded. Each subject will participate in both residual limb shape capture methods during the first study visit (order randomly assigned), but only one study socket (either the study helper assisted socket with digital methods, or the prosthetist made socket with traditional methods) will be used for outcomes testing (randomly assigned and blinded to the participant).
  Care Provider: The prosthetist will fabricate the prosthetist socket using traditional methods, thereby knowing study socket and participant randomization. However, the investigators will apply apply a fabric cover to the sockets (both sensorized as-prescribed and study sockets) during visits 3 and 4. This method blinds the prosthetist during the distal end residual limb pressure measurements.
  Outcomes Assessor. The study staff collecting patient reported outcomes will also be blinded, as they will not know which socket the participant received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caregiver socket (Experimental): Participants will wear a prosthetic socket whose shape was captured by a study helper using digital methods (i.e., a 3D scanner).
  Interventions: Device: Caregiver socket
- Prosthetist socket (Experimental): Participants will wear a prosthetic socket whose shape was captured by a prosthetist using traditional, hand casting methods.
  Interventions: Device: Prosthetist socket

INTERVENTIONS:
Device: Caregiver socket — A prosthetic socket whose shape was captured by a study helper using digital methods (i.e., 3D scanner). The digital file describing the socket dimensions will be sent to a central fabrication facility where the prosthetic socket will be manufactured.
  Arms: Caregiver socket
Device: Prosthetist socket — A prosthetic socket whose shape was captured by a prosthetist using traditional, hand casting methods. The hand cast will be plaster filled to create a positive model. A prosthetist socket will be fabricated over the positive model using thermoplastic materials.
  Arms: Prosthetist socket

SUMMARY:
When the prosthetic socket of a Veteran with a lower limb amputation no longer fits or is damaged beyond repair, a new prosthetic socket is warranted. The provision of a new socket requires multiple clinical visits which can place a high travel burden and potential pandemic exposure stress on Veterans who live in rural communities far from VA Medical Centers or alternative prosthetic clinics. This research seeks to determine if one of the in-person visits traditionally needed to obtain a well-fitting prosthesis can be performed remotely with the assistance of a helper. The investigators seek to discover if an untrained individual (a helper) can wield inexpensive, easy to use, digital technology to capture the shape of a residual limb to see if it can be used to fabricate a prosthetic socket that fits at least as well as one fabricated by a prosthetist using traditional, hand casting methods in the clinic.

The expected result of this research is an evidence-based prosthetic fabrication process that reduces Veteran travel burden while providing a prosthesis that fits at least as well as the current standard-of-care. The upshot is a clear improvement in prosthetic provision for Veterans, particularly for those who live in rural communities.

To make this determination, the investigators will perform a between-subject experiment with two specific aims. To determine differences in goodness of fit between the two study sockets, the investigators will use both patient reported outcomes, and measurements of the pressure applied to the distal end of the residual limb.

Specific Aim 1: Determine if patient reported outcomes, by subjects wearing a prosthetic socket whose shape was captured with study helper assistance, are at least as good as those reported by subjects wearing a socket whose shape was captured by a prosthetist. The investigators propose to recruit Veterans with a below knee amputation and their study helpers to participate in a human subject experiment. Participants will be randomly assigned and fit with either a prosthesis made with study helper assistance and digital methods, or one made wholly by a prosthetist using traditional methods. Patient reported outcome metrics will be collected while the subject is still wearing their as-prescribed socket at the beginning of the study (baseline), and again after wearing the study prosthesis for two weeks.

Specific Aim 2: Determine if distal end residual limb pressure, measured from a group of individuals fit with a prosthetic socket whose shape was captured with study helper assistance using digital methods, are no worse than those measured from a group of individuals fit with a prosthetic socket whose shape was captured by a prosthetist using traditional methods. Concurrent with the human subject procedures briefly described above, the investigators propose to fabricate duplicates (copies) of the two prosthetic sockets used by each subject in Specific Aim 1. A novel sensor will be embedded in these duplicate sockets which can measure the pressure applied to the distal end of the residual limb. Measurements of distal end residual limb pressure while standing and walking for both the as-prescribed and study sockets will be collected at the beginning of the study (baseline), and again after two weeks.

The data from the investigators' experiments will be used to determine if residual limb shape capture by a helper using digital technologies can be used to make prosthetic sockets that fit at least as well as those made by a prosthetist using traditional, hand casting techniques.

One third of all Veterans live in rural communities far from VA Medical Centers. When Veterans with a lower limb amputation need a new prosthetic socket, attending in-person clinical visits can be a challenge. If the hypotheses are supported, this research will provide evidence to support the use of digital technology as part of clinical practice, enabling a remote, study helper enabled alternative to one of the in-person clinical visits needed to fabricate a well-fitting prosthesis.

DETAILED DESCRIPTION:
The objective of this research is to determine if advances in technology, namely digital methods to capture residual limb shape, can meet the well-fitting prosthetic socket standard-of-care with the added benefits of improved access and service delivery. The current standard of care for prosthetic provision requires multiple, in-person clinical visits between the Veteran and their prosthetist. Separate visits for residual limb shape capture, check socket fitting, and definitive socket delivery are required every time a new socket is needed. For Veterans who live in rural communities far from VA facilities, the challenges associated with attending these clinical visits can be a significant burden. This research seeks to determine if the residual limb shape capture visit can be performed remotely with the assistance of a study helper using digital methods.

Of paramount concern when providing a prosthesis to a Veteran with a lower limb amputation is obtaining a good fit. Prosthetic sockets that fit poorly are either worn sparingly or not at all. Obtaining a good fit is a process. Veterans know it when they wear a well-fitting prosthesis and prosthetists know it when they see it (lack of reactive hyperemia). Patient reported outcomes play an important role whereby the prosthetist solicits feedback from the patient about how the check socket feels and the location of any perceived discomfort. This informal approach is infrequently supplemented with qualitative survey instruments. Reducing or eliminating excessive distal end pressure is also essential as the distal end tissues of the residual limb can rarely support body weight loads without discomfort or injury. However, no instrument to directly measure distal end residual limb pressures is commercially available.

The investigators propose to determine if a prosthetic socket, whose shape is captured remotely by a study helper using a digital scanner, fits at least as well as a prosthetic socket whose shape is captured in-person by a prosthetist using traditional hand casting methods. If it does, then rural Veterans with a helper could forgo a clinical visit. To make this determination, the investigators propose to perform a between-subject experiment with two specific aims.

Specific Aim 1: Determine if patient reported outcomes, reported by a group of individuals fit with a prosthetic socket whose shape was captured with study helper assistance using digital methods, are at least as good as those reported by a different group of individuals fit with a prosthetic socket whose shape was captured by a prosthetist using traditional methods. The investigators propose to recruit ambulatory Veterans with unilateral transtibial amputation (n=20) and their study helpers (n=20) to participate in a between-subject experiment. Participants will be randomly assigned and fit with either a prosthesis made with study helper assistance and digital methods, or one made wholly by a prosthetist using traditional methods. Patient reported outcome metrics will be collected while the subject is still wearing their as-prescribed socket (baseline) at the beginning of the study, and again after wearing the study prosthesis for two weeks.

Specific Aim 2: Determine if distal end residual limb pressure, measured from a group of individuals fit with a prosthetic socket whose shape was captured with study helper assistance using digital methods, are no worse than those measured from a group of individuals fit with a prosthetic socket whose shape was captured by a prosthetist using traditional methods. In addition to the human subject procedures of Specific Aim 1, the investigators further propose to fabricate two duplicate prosthetic sockets for each subject: one duplicate of the subject's as-prescribed socket and one duplicate of the study socket randomly assigned to the subject in Specific Aim 1. Embedded in the distal end of these duplicate sockets will be a novel pressure sensor. Distal end residual limb pressure while standing and walking will be measured while the subject is still wearing their as-prescribed socket (baseline), and again after wearing the study prosthesis for two weeks.

The proposed research will discover if it is possible to forgo one of the clinical visits needed to fabricate a well-fitting prosthesis. It is the investigators' hope that this research will advance the use of technology in the provisioning of prostheses, particularly to Veterans who live in rural communities far from VA Medical Centers or alternative service providers.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* Been fit with a prosthesis and used it for at least 6 months
* Wear the prosthesis for 4 or more hours on average per day
* Has a prosthesis that bolts to the bottom of the socket
* Be at least one-year post-amputation
* Able to walk on a treadmill
* Have an eligible and available study helper

Exclusion Criteria:

* Improper fit and suspension with current prosthesis and one cannot be achieved with clinical resources
* Current skin irritation or injury on residual limb
* Osteoarthritis, injury, or pain that interferes with walking ability
* Currently incarcerated
* Pregnant
* Inadequate cognitive function or language proficiency to consent to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Socket Comfort Score (SCS) | After a two week acclimation period where the participant wears the study prosthesis in the home, community, and work environments.
  Participants rate the comfort of their socket on an 11-point scale where 0 and 10 represent the most uncomfortable and the most comfortable socket imaginable, respectively.
Comprehensive Lower-limb Amputee Socket Survey (CLASS) Stability Score | After a two week acclimation period where the participant wears the study prosthesis in the home, community, and work environments.
  Participants rate their stability when wearing their prosthesis on a 4-point scale where 1 indicates they strongly disagree and 4 indicates they strongly agree that they feel stable and balanced in their socket when they are sitting, standing, walking, or ascending/descending stairs. The Stability score is reported as a percentage of awarded score / total possible score.
Comprehensive Lower-limb Amputee Socket Survey (CLASS) Suspension Score | After a two week acclimation period where the participant wears the study prosthesis in the home, community, and work environments.
  Participants rate their security with their prosthetic suspension on a 4-point scale where 1 indicates they strongly disagree and 4 indicates they strongly agree that they feel secure in their socket with no excessive movement when they are sitting, standing, walking, or ascending/descending stairs. The Suspension score is reported as a percentage of awarded score / total possible score.
Comprehensive Lower-limb Amputee Socket Survey (CLASS) Comfort Score | After a two week acclimation period where the participant wears the study prosthesis in the home, community, and work environments.
  Participants rate their comfort when wearing their prosthesis on a 4-point scale where 1 indicates they strongly disagree and 4 indicates they strongly agree that they feel comfortable in their socket when they are sitting, standing, walking, or ascending/descending stairs. The Comfort score is reported as a percentage of awarded score / total possible score.
Standing distal end residual pressure | After a two week acclimation period where the participant wears the study prosthesis in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant stands for 60 seconds. The first and last fifteen seconds of the standing pressure data (60 second trial) will be truncated and the mean pressure will be calculated from the middle 30 seconds of each trial (3 repeated trials).
Walking distal end residual limb pressure | After a two week acclimation period where the participant wears the study prosthesis in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant walks on a treadmill at their self-selected speed for 60 seconds. The first and last fifteen seconds of the walking pressure data (60 second trial) will be truncated and the mean pressure will be calculated from the middle 30 seconds of each trial (3 repeated trials).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A de-identified, anonymized dataset will be created and available to the public via a VA authorized website. Where possible, the investigators will work with manuscript publishers to link the final study data sets as an appendix to published manuscripts. By providing de-identified datasets in open file formats (e.g., .txt, .xls, .mat) along with clearly documented instructions for processing, interested recipients will be able to reproduce and build on the same techniques which the investigators will outline in our publications. A public release identifier for each subject's data (e.g., CGS_001, CGS_002) will be created and randomly paired with de-identified study data. Data will consist of subject demographics, test, and questionnaire results. There will be no tractable way to re-match these data to the subject. Our methods will be verified by the VAPSHCS Privacy Officer.
Time Frame: Within six months of publication of final study findings.
Access Criteria: Open access through PubMed Central, SimTK, PhysioNet, or other similar open-source data repository websites.